CLINICAL TRIAL: NCT03700853
Title: Validity And Reliability Of A Dysphagia Trained Nurse Assessment (DTNAx) Tool In Acute Stroke
Brief Title: Validation and Reliability Testing of Dysphagia Trained Nurse Assessment
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17027
Record Dates: First submitted 2018-09-24; First posted 2018-10-09 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Dysphagia Following Cerebral Infarction; Dysphagia Following Nontraumatic Intracerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dysphagia Trained Nurse Assessment (DTNAx) — Bedside swallowing assessment carried out by trained nurses

SUMMARY:
Nurses at Royal Derby Hospital, UK have been trained to use a comprehensive protocol based dysphagia assessment (Dysphagia Trained Nurse Assessment (DTNAx)) to assess all acute stroke patients on admission. This study aims to validate the tool by comparing it to the gold standard assessment - Videofluoroscopy and usual assessment by a Speech and Language Therapist. Inter-rater and intra-rater reliability will also be tested by comparing the assessment results of two different nurses or the same nurse.

DETAILED DESCRIPTION:
Speech and Language Therapists (SLTs) at Royal Derby Hospital (RDH) have developed a tool that trained nurses can use to carry out swallowing assessments with patients following a stroke. It consists of checks to ensure the patient is alert/well enough, checks any abnormalities in the muscles of the mouth or throat and trials different types of foods/drinks. If they 'pass' the assessment patients are started with regular diet and fluids. If they have dysphagia the nurses can recommend modified foods/drinks if they have found to be safe during the assessment. If the patients 'fail' with all trials - they remain nil by mouth. Around 50% of patients who have a stroke have difficulties swallowing (dysphagia). If dysphagia is identified early it reduces secondary complications such as pneumonia. There are no similar tools in the UK that have been tested to check they are doing what they say they are doing (validity) or the results are the same no matter which trained nurse uses the tool (reliability). This study aims to test the validity and reliability of the Dysphagia Trained Nurse Assessment DTNAx that is currently used in the acute stroke pathway at RDH.

Over an 18 month period we aim to recruit 50 patients admitted to RDH with a new stroke and who have had an initial DTNAx. The results of the DTNAx will be compared to the gold standard dysphagia assessment - videofluoroscopy - a video xray of swallowing and also compared to the usual SLT assessment. We can calculate whether the tool identifies dysphagia and whether the recommendations made by using the tool are accurate and safe. To test reliability - the DTNAx will be repeated by the same nurse or by a different nurse. The patients will be involved in the study for approximately 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18
* Clinical diagnosis of stroke (ischaemic or haemorrhagic)

Exclusion Criteria:

* Dysphagia of another cause
* Unable to tolerate VFS due to agitation or severe cognitive difficulties (patients need to be able to sit in a suitable chair - REA assist, 9L, Mangar Porter, Tilt and Space etc. for VFS)
* Not medically well enough to undertake assessments (as determined by the clinical care team)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 who have been admitted to the Acute Stroke Unit who have a clinical diagnosis of stroke, who have had a DTNAx. They are medically stable, able to sit out in a suitable chair and have no previous dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Evidence of dysphagia on gold standard test | 24 hours
  Cut off scores as per Standardised and reliability assessment: Modified Barium Swallow Impairment Profile on Videofluoroscopy assessment
Fluid Recommendation on gold standard test | 24 hours
  On Videofluoroscopy - Least restrictive fluid with Penetration Aspiration Scale of 1 or 2, MBSImP pharyngeal residue rating of <3, number of swallows < 3.
Diet Recommendation on gold standard test | 24 hours
  On Videofluoroscopy - Least restrictive fluid with Penetration Aspiration Scale of 1 or 2, MBSImP pharyngeal residue rating of <3, number of swallows < 3. • If solid bolus trialled (forkmashable/normal) - mastication needs to be timely and complete - therefore MBS-Imp score on Component 3 Bolus preparation/mastication = 0

SECONDARY OUTCOMES:
Outcome of SLT clinical bedside assessment (SLTAx) | 24 hours
  This is not a standardised test - but it is usual practice. Information will be collected on the subtest carried out in the assessment. Ultimately the outcomes that are measured are SLT judgement of: presence of dysphagia, safe diet recommendation, safe fluid recommendation
Outcome of 2nd Dysphagia Trained Nurse Assessment (DTNAx) | 24 hours
  The DTNAx standardised assessment and is the assessment that is being validated in this study. To measure intra and inter rater reliability this outcome measure is the outcome of a second DTNAx assessment - specifically the safe diet recommendation and safe fluid recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy England, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided